CLINICAL TRIAL: NCT01826786
Title: The Effects of JNJ-42165279 on the Neural Basis of Anxiety Disorders in Healthy Male Subjects
Brief Title: The Effects of JNJ-42165279 on the Neural Basis of Anxiety Disorders in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CR100975; 42165279ANX1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: Healthy; Anxiety Disorders; Anxiety Modulation; Male
MeSH Terms: conditions — Anxiety Disorders | interventions — JNJ-42165279

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- JNJ-42165279 (100 mg) (Experimental)
  Interventions: Drug: JNJ-42165279 (100 mg)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-42165279 (100 mg) — JNJ-42165279 (100 mg/day) will be orally administered once daily for 4 consecutive days.
  Arms: JNJ-42165279 (100 mg)
Drug: Placebo — Matching placebo to JNJ-42165279 will be orally administered once daily for 4 consecutive days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the potential efficacy of JNJ-42165279 in treating anxiety disorders through evaluation of brain activation patterns using imaging technology in healthy volunteers.

DETAILED DESCRIPTION:
This is a single site, double-blind (neither investigator nor the participant knows the treatment that the participant receives) study. The study will consist of a screening phase (1-2 visits), a treatment phase (4 visits), and a post treatment phase (follow-up safety visit, 7 to 14 days after the last dose of the study drug). During the screening phase, participants will be evaluated to determine if they meet the study eligibility criteria, which will include collection of blood and urine samples. During the treatment phase, eligible participants will be assigned by chance (like a toss of a coin) to receive either JNJ-42165279 100 mg or placebo once daily during 4 consecutive visits to the clinic. Placebo is an inactive substance that is compared with a drug to test whether the drug has a real effect. The potential of the drug to treat anxiety will be assessed on Day 4 of the treatment phase. The primary assessment, Blood Oxygen Level Dependent Functional Magnetic Resonance Imaging (BOLD-fMRI), will measure brain activity patterns while participants complete 3 emotionally-provoking tasks. Additionally, participants' startle responses (eye blinks) will be evaluated in two emotionally-provoking behavioral tasks outside of the scanner. Questionnaires will be completed to evaluate participants' mood, and blood samples will be collected to measure concentrations of JNJ-42165279 and biomarkers of drug activity.

Safety will be monitored throughout the study, including adverse events, vital signs (blood pressure and heart rate), 12-lead ECGs, physical examinations, clinical safety laboratories, evaluation of suicidal risk, and a Walk and Turn test. The total study duration will be approximately 46 days.

ELIGIBILITY:
Inclusion criteria

* Good general health
* Body mass index between 18 and 30 kg/m2 and body weight not less than 50 kg
* Must adhere to required contraception during and for 3 months after study
* Must agree to not donate sperm during and for 3 months after study
* Must agree to not donate blood during and for 1 month after study
* Able to speak and understand English fluently

Exclusion criteria:

* Clinically significant medical or psychiatric illness
* Any contraindication to magnetic resonance imaging
* Unable to pass hearing test
* Alcohol or substance abuse; excessive nicotine or caffeine use
* Recently received an investigational drug, vaccine, or invasive medical device
* Unable to abide by protocol restrictions on use of other medications

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Brain activity patterns in the amygdala (almond-shaped part of the brain associated with motivation and emotional behavior) | Day 4
  BOLD-fMRI percent signal changes during an Emotional Face Processing task.

SECONDARY OUTCOMES:
Brain activity patterns in multiple areas of the emotional brain neurocircuitry | Day 4
  BOLD-fMRI percent signal changes during emotionally-provoking tasks (pictures of emotional faces, periods of breathing restriction, presentations of a loud noise).
Startle response | Day 4
  Eye blink responses to a loud noise during 2 emotionally-provoking tasks outside of the MRI scanner.
The number of volunteers who experience adverse events as a measure of safety and tolerability. | Day -28 to Day 18

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- La Jolla, California, United States